CLINICAL TRIAL: NCT04870580
Title: [18F] FDOPA PET Imaging in Glioma: Feasibility Study for PET Guided Brain Biopsy
Acronym: FIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127427; 272494 (Other: IRAS)
Record Dates: First submitted 2021-04-12; First posted 2021-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): PET/CT with fluorodopa tracer
  Interventions: Diagnostic Test: Fluorodopa PET tracer

INTERVENTIONS:
Diagnostic Test: Fluorodopa PET tracer — PET/CT scan using fluorodopa tracer

SUMMARY:
[18F]fluorodopa (3, 4-dihydroxy-6-[18F]fluoro-L-phenylalanine/ FDOPA) is an amino acid PET tracer originally developed for brain imaging in patients with movement disorders but has been found to be useful in brain tumour imaging. [18F]fluorodopa has been demonstrated to be predominantly transported by the L-type amino acid transporter without significant uptake into surrounding normal brain parenchyma with the exception of the basal ganglia. Assessing the feasibility of performing PET guided histopathology in a single and multi-site setting will be crucial in order to use PET as a planning tool for brain biopsy to detect high-grade transformation in low-grade gliomas.

DETAILED DESCRIPTION:
Glioma is a cancer of unmet need, where survival trends have not significantly changed for decades. The distinction between high-grade (HGG) and low-grade glioma (LGG) is important as both entities confer different prognoses and management strategies. This distinction is normally made on biopsy sampling and conventional imaging. However, sampling errors are not uncommon due to the heterogeneous nature of glioma. Case series have described under-grading of gliomas on biopsy in 28% to 63% of cases. Furthermore, up to one third of high-grade gliomas may not display the typical imaging characteristics (enhancement) of a high-grade glioma. Therefore, more accurate imaging may help to make this distinction and guide biopsy and clinical management decisions at the outset.

There has been growing interest in the use of amino acid PET in glioma imaging. Transport of amino acids across the blood brain barrier and low physiological levels of tracer uptake within the brain allow for good tumour visualisation. The most frequently used amino acid PET tracers described in clinical literature are [11C]methionine, [18F]fluoroethyltyrosine and [18F]fluorodopa, which predominantly reflect leucine transport, being mainly transported by LAT1, a high affinity leucine transporter. Alongside depiction of tumour volume, described roles of amino acid PET include differentiation of true disease progression from pseudo progression, detection of residual disease in the post-surgical patient, biopsy guidance and prognostication.

Rationale The primary objective of the study will be to establish the feasibility of performing [18F]fluorodopa PET guided histopathology in a single and multi-site setting. Basic tumour characterisation (for example Ki67 expression and detection of IDH mutations) will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Diagnosed with low-grade glioma based on clinical standard of care imaging and scheduled for primary surgical resection of low-grade glioma
3. Females of childbearing potential and males agree to use an effective method of contraception from the time consent is signed until 1 week after surgery.
4. Females of childbearing potential have a negative urine pregnancy test within 7 days prior to being registered. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
5. Willing and able to provide written informed consent

Exclusion Criteria:

1. Females who are pregnant, planning pregnancy or breastfeeding
2. Concurrent and/or recent involvement in other research or use of another experimental investigational medicinal product that is likely to interfere with the study medication within 28 days of study enrolment.
3. MRI contraindicated (e.g. implanted electric and electronic devices, heart pacemakers, insulin pumps, implanted hearing aids, neurostimulators, intracranial metal clips, metallic bodies in the eye).
4. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor study candidate or could interfere with protocol compliance or the interpretation of study results.
5. Neoadjuvant chemotherapy/radiotherapy treatment for low-grade glioma which would interfere with the interpretation of study results.
6. Any other problems that may make the patient unable to tolerate the PET scans (e.g. claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of PET guided histopathology in a single and multi-site setting. | 2 years
  Assessment of tumour standardised uptake values (SUV) from [18F]fluorodopa PET with matched histopathology data from biopsies for evaluable patients from a single site and multiple sites. The percentage of cases where it is possible to collect this data will inform the feasibility of performing the assessments in a single-site and multi-site setting with a 70% threshold used to determine feasibility.

SECONDARY OUTCOMES:
To investigate the inter-observer variation (IOV) in tumour to background uptake measurements to assess reliability. | 2 years
  IOV in tumour to background uptake measurements
To characterise dopamine uptake in high-grade glioma and low-grade glioma. | 2 years
  SUV/TBR corresponding to the optimal cut-off value for high-grade and low-grade glioma on receiver operating characteristic curve analysis.
To provide data on the proportion of high-grade transformation in low-grade glioma. | 2 years
  Proportion of patients showing high-grade transformation following histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Higgins, Principal Investigator — University College, London
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No